CLINICAL TRIAL: NCT02003209
Title: A Randomized Phase III Trial Evaluating Pathologic Complete Response Rates in Patients With Hormone Receptor-Positive, HER2-Positive, Large Operable and Locally Advanced Breast Cancer Treated With Neoadjuvant Therapy of Docetaxel, Carboplatin, Trastuzumab, and Pertuzumab (TCHP) With or Without Estrogen Deprivation
Brief Title: Docetaxel, Carboplatin, Trastuzumab, and Pertuzumab With or Without Estrogen Deprivation in Treating Patients With Hormone Receptor-Positive, HER2-Positive Operable or Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-02228; NCI-2013-02228 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NSABP-B-52 (Other: NRG Oncology); NSABP-B-52 (Other: CTEP); U10CA012027 (NIH); U10CA180868 (NIH)
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Results first posted 2023-06-12 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: HER2-Positive Breast Carcinoma; Hormone Receptor-Positive Breast Carcinoma; Stage IB Breast Cancer AJCC v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Aromatase Inhibitors; Carboplatin; Docetaxel; Goserelin; pertuzumab; 2C4 antibody; Trastuzumab; CT-P6; PF-05280014; trastuzumab biosimilar HLX02; Ogivri; Ontruzant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (combination chemotherapy, surgery, radiation) (Active Comparator): NEOADJUVANT: Patients receive docetaxel IV over 60 minutes, carboplatin IV over 30-60 minutes, trastuzumab IV over 30-90 minutes, and pertuzumab IV over 30-60 on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients enrolled after Amendment #4 undergo 2 core biopsies prior to course 3 of treatment.
  SURGERY: Patients undergo lumpectomy or mastectomy.
  RADIATION: Patients undergo whole breast irradiation within 8 weeks following surgery.
  ADJUVANT: Patients receive trastuzumab IV over 30-60 minutes every 21 days for up to 1 year.
  Interventions: Drug: Carboplatin; Other: Cytology Specimen Collection Procedure; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Biological: Pertuzumab; Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery; Biological: Trastuzumab; Radiation: Whole Breast Irradiation
- Arm II (chemo, estrogen deprivation, surgery, radiation) (Experimental): NEOADJUVANT: All patients receive docetaxel, carboplatin, trastuzumab, and pertuzumab as in arm I. Premenopausal patients also receive goserelin acetate SC every 28 days until surgery and aromatase inhibition therapy at the investigator's discretion daily until 1 day before surgery. Postmenopausal patients receive aromatase inhibition therapy at the investigator's discretion daily until 1 day before surgery. Patients enrolled after Amendment #4 undergo 2 core biopsies prior to course 3 of treatment.
  SURGERY: Patients undergo lumpectomy or mastectomy.
  RADIATION: Patients undergo whole breast irradiation within 8 weeks following surgery.
  ADJUVANT: Patients receive trastuzumab IV over 30-60 minutes every 21 days for up to 1 year.
  Interventions: Drug: Aromatase Inhibition Therapy; Drug: Carboplatin; Other: Cytology Specimen Collection Procedure; Drug: Docetaxel; Drug: Goserelin Acetate; Other: Laboratory Biomarker Analysis; Biological: Pertuzumab; Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery; Biological: Trastuzumab; Radiation: Whole Breast Irradiation

INTERVENTIONS:
Drug: Aromatase Inhibition Therapy — Given at the investigator's discretion
  Other Names: Aromatase Inhibition
  Arms: Arm II (chemo, estrogen deprivation, surgery, radiation)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Cytology Specimen Collection Procedure — Undergo 2 core biopsies
  Other Names: Cytologic Sampling
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
  Arms: Arm II (chemo, estrogen deprivation, surgery, radiation)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pertuzumab — Given IV
  Other Names: 2C4; 2C4 Antibody; BCD-178; EG1206A; HLX11; HS627; MoAb 2C4; Monoclonal Antibody 2C4; Omnitarg; Perjeta; Pertuzumab Biosimilar BCD-178; Pertuzumab Biosimilar EG1206A; Pertuzumab Biosimilar HLX11; Pertuzumab Biosimilar HS627; Pertuzumab Biosimilar TQB2440; Rhumab 2C4; rhuMAb2C4; RO4368451; TQB 2440; TQB-2440; TQB2440
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Therapeutic Conventional Surgery — Undergo lumpectomy or mastectomy
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Biceltis; CANMab; CT-P06; CT-P6; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Hercessi; Herclon; Hertraz; Herwenda; Herzuma; HLX 02; HLX-02; HLX02; Kanjinti; Ogivri; Ontruzant; PF 05280014; PF-05280014; PF05280014; QL 1701; QL-1701; QL1701; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; Trastuzumab Biosimilar CT-P6; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar QL1701; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-herw; Trastuzumab-pkrb; Trastuzumab-qyyp; Trastuzumab-strf; Trastuzumab-zerc; Trazimera; Zercepac
Radiation: Whole Breast Irradiation — Undergo whole breast irradiation

SUMMARY:
This randomized phase III trial studies docetaxel, carboplatin, trastuzumab, and pertuzumab with estrogen deprivation to see how they work compared to docetaxel, carboplatin, trastuzumab, and pertuzumab without estrogen deprivation in treating patients with hormone receptor-positive, human epidermal growth factor receptor 2 (HER2)-positive breast cancer that is operable or has spread from where it started to nearby tissue or lymph nodes (locally advanced). Drugs used in chemotherapy, such as docetaxel, carboplatin, trastuzumab, and pertuzumab, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Estrogen can cause the growth of breast cancer cells. Hormone therapy using goserelin acetate and aromatase inhibition therapy may fight breast cancer by blocking the use of estrogen by the tumor cells. Radiation therapy uses high energy x rays to kill tumor cells. Giving combination chemotherapy and radiation therapy with or without hormone therapy may be an effective treatment for hormone receptor-positive, HER2-positive, operable or locally advanced breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the addition of estrogen deprivation to neoadjuvant therapy consisting of therapy of docetaxel, carboplatin, trastuzumab, and pertuzumab (TCHP) yields a greater rate of pathologic complete response (pCR) (breast and nodes) than TCHP alone when administered to women with operable, hormone receptor-positive, HER2-positive breast cancer.

SECONDARY OBJECTIVES:

I. To determine whether the addition of estrogen deprivation to neoadjuvant therapy consisting of TCHP will increase the pCR rate in the breast compared to TCHP alone when administered to women with operable, hormone receptor-positive, HER2-positive breast cancer.

II. To determine whether the addition of estrogen deprivation to neoadjuvant therapy consisting of TCHP improves recurrence-free interval (RFI) in women with operable, hormone receptor-positive, HER2-positive breast cancer.

III. To determine whether the addition of estrogen deprivation to neoadjuvant therapy consisting of TCHP improves overall survival (OS) in women with operable, hormone receptor-positive, HER2-positive breast cancer.

IV. To compare the rates of second primary invasive cancer by treatment arm. V. Assessment of patterns of pCR, RFI, and OS by menopausal status. VI. To evaluate the cardiac toxicity associated with each of the regimens. VII. To compare the effect of adding estrogen deprivation to neoadjuvant therapy on endocrine-related symptoms in all patients by treatment arm.

VIII. To compare the effect of adding estrogen deprivation to neoadjuvant therapy on vasomotor symptoms, musculoskeletal, and vaginal complaints as well as quality of life.

IX. To determine a relationship between pCR and a potential mechanism of resistance/sensitivity in hormone receptor-positive, HER2-positive tumors.

X. To evaluate tumor infiltrating lymphocytes (TILs) and immune biomarkers as predictors of pCR.

XI. To study early changes in TILs and other immune biomarkers in response to TCHP.

OUTLINE: Patients are randomized to 1 of 2 treatments arms.

NEOADJUVANT:

ARM I: Patients receive docetaxel intravenously (IV) over 60 minutes, carboplatin IV over 30-60 minutes, trastuzumab IV over 30-90 minutes, and pertuzumab IV over 30-60 on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients enrolled after Amendment #4 undergo 2 core biopsies prior to course 3 of treatment.

ARM II: All patients receive docetaxel, carboplatin, trastuzumab, and pertuzumab as in arm I. Premenopausal patients also receive goserelin acetate subcutaneously (SC) every 28 days until surgery and aromatase inhibition therapy at the investigator's discretion daily until 1 day before surgery. Postmenopausal patients receive aromatase inhibition therapy at the investigator's discretion daily until 1 day before surgery. Patients enrolled after Amendment #4 undergo 2 core biopsies prior to course 3 of treatment.

SURGERY: Patients undergo lumpectomy or mastectomy.

RADIATION: Patients undergo whole breast irradiation within 8 weeks following surgery.

ADJUVANT: Patients receive trastuzumab IV over 30-60 minutes every 21 days for up to 1 year.

After completion of study treatment, patients are followed up every 6, 9, 12, and 18 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a life expectancy of at least 10 years, excluding their diagnosis of breast cancer; (comorbid conditions should be taken into consideration, but not the diagnosis of breast cancer)
* Women of reproductive potential must agree to use an effective non-hormonal method of contraception during study therapy (chemotherapy, trastuzumab, pertuzumab, and estrogen deprivation therapy) and for at least 7 months after the last dose of study therapy
* Submission of tumor samples is required for all patients; the local pathology department policy regarding release of tumor samples must be considered in the screening process; patients whose tumor samples are located in a pathology department that by policy will not submit any samples for research purposes should not be approached for participation in the B-52 trial
* The patient must have signed and dated an Institutional Review Board (IRB)-approved consent form that conforms to federal and institutional guidelines
* The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Clinical staging for the primary tumor can be cT1c (must be 2.0 cm) or T2-T4 if clinically node negative; if the regional lymph nodes are cN1 and cytologically or histologically positive or if cN2-N3 with or without a biopsy, the primary breast tumor can be cT0-T4
* The diagnosis of invasive adenocarcinoma of the breast must have been made by core needle biopsy
* Ipsilateral axillary lymph nodes must be evaluated by imaging (mammogram, ultrasound, and/or magnetic resonance imaging [MRI]) within 6 weeks prior to randomization; if suspicious or abnormal, fine needle aspirate (FNA) or core biopsy is recommended, also within 6 weeks prior to randomization; findings of these evaluations will be used to determine the nodal status prior to randomization:

  * Nodal status - negative

    * Imaging of the axilla is negative
    * Imaging is suspicious or abnormal but the FNA or core biopsy of the questionable node(s) on imaging is negative
  * Nodal status - positive

    * FNA or core biopsy of the node(s) is cytologically or histologically suspicious or positive
    * Imaging is suspicious or abnormal but FNA or core biopsy was not performed
* Patients may be premenopausal or postmenopausal at the time of randomization; for study purposes, postmenopausal is defined as:

  * Age 56 or older with no spontaneous menses for at least 12 months prior to study entry; or
  * Age 55 or younger with no spontaneous menses for at least 12 months prior to study entry (e.g., spontaneous or secondary to hysterectomy) and with a documented estradiol level in the postmenopausal range according to local institutional/laboratory standard; or
  * Documented bilateral oophorectomy
* The tumor must have been determined to be HER2-postive as follows:

  * Immunohistochemistry (IHC) 3+ or
  * In situ hybridization (ISH)-positive (defined by ratio of HER2 to circulating endothelial progenitors [CEP]17 >= 2.0 or HER2 gene copy number >= 6 per nucleus)
* The tumor must have been determined to be estrogen receptor (ER) and/or progesterone (PgR) positive assessed by current American Society of Clinical Oncology (ASCO)/College of American Pathologist (CAP) guideline recommendations for hormone receptor testing; patients with >= 1% ER or PgR staining by IHC are considered positive
* Absolute neutrophil count (ANC) must be >= 1200/mm^3
* Platelet count must be >= 100,000/mm^3
* Hemoglobin must be >= 10 g/dL
* Total bilirubin must be =< upper limit of normal (ULN) for the lab unless the patient has a bilirubin elevation > ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin
* Alkaline phosphatase must be =< 2.5 x ULN for the lab
* Aspartate aminotransferase (AST) must be =< 1.5 x ULN for the lab
* Alkaline phosphatase and AST may not both be > the ULN; for example, if the alkaline phosphatase is > the ULN but =< 2.5 x ULN, the AST must be =< the ULN; if the AST is > the ULN but =< 1.5 x ULN, the alkaline phosphatase must be =< ULN; Note: If alanine aminotransferase (ALT) is performed instead of AST (per institution's standard practice), the ALT value must be =< 1.5 x ULN; if both were performed, the AST must be =< 1.5 x ULN
* Patients with AST or alkaline phosphatase > ULN are eligible for inclusion in the study if liver imaging (computed tomography [CT], MRI, positron emission tomography [PET]-CT, or PET scan) performed within 6 weeks prior to randomization does not demonstrate metastatic disease and the requirements are met
* Patients with alkaline phosphatase that is > ULN but =< 2.5 x ULN or unexplained bone pain are eligible for inclusion in the study if a bone scan, PET-CT scan, or PET scan performed within 6 weeks prior to randomization does not demonstrate metastatic disease
* Within 6 weeks prior to randomization, the most recent serum creatinine must be =< ULN or measured or calculated creatinine clearance must be > 60 mL/min
* Left ventricular ejection fraction (LVEF) assessment must be performed within 90 days prior to randomization; (LVEF assessment performed by 2-dimensional [2-D] echocardiogram is preferred; however, multi gated acquisition scan [MUGA] scan may be substituted based on institutional preferences); the LVEF must be >= 50% regardless of the cardiac imaging facility's lower limit of normal; note: since the pre-entry LVEF serves as the baseline for comparing subsequent LVEF assessments, it is critical that this baseline study be an accurate assessment; if the baseline LVEF is > 65%, the investigator is encouraged to have the accuracy of the initial LVEF result confirmed and repeat the test if the accuracy is uncertain

Exclusion Criteria:

* FNA alone to diagnose the breast cancer
* Excisional biopsy or lumpectomy performed prior to randomization
* Surgical axillary staging procedure prior to randomization; pre-neoadjuvant therapy sentinel node biopsy is not permitted
* Definitive clinical or radiologic evidence of metastatic disease; (chest imaging [mandatory for all patients] and other imaging [if required] must have been performed within 90 days prior to randomization)
* Synchronous bilateral invasive breast cancer
* Synchronous or previous contralateral invasive breast cancer; (patients with synchronous and/or previous contralateral ductal carcinoma in situ [DCIS] or lobular carcinoma in situ [LCIS] are eligible)
* Any previous history of ipsilateral invasive breast cancer or ipsilateral DCIS; (patients with synchronous or previous ipsilateral LCIS are eligible)
* Treatment including radiation therapy (RT), chemotherapy, targeted therapy, or endocrine therapy for the currently diagnosed breast cancer prior to randomization
* Previous endocrine therapy such as raloxifene or tamoxifen (or other selective estrogen receptor modulator [SERM]) or an aromatase inhibitor for any malignancy
* Previous therapy with anthracycline, taxanes, carboplatin, trastuzumab, or other HER2 targeted therapies for any malignancy
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormone replacement therapy, etc. (these patients are eligible if this therapy is discontinued prior to randomization)
* History of non-breast malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 5 years prior to randomization
* Cardiac disease (history of and/or active disease) that would preclude the use of the drugs included in the treatment regimens; this includes but is not confined to:

  * Active cardiac disease:

    * Angina pectoris that requires the use of anti-anginal medication;
    * Ventricular arrhythmias except for benign premature ventricular contractions;
    * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication;
    * Conduction abnormality requiring a pacemaker;
    * Valvular disease with documented compromise in cardiac function; and
    * Symptomatic pericarditis
  * History of cardiac disease:

    * Myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular (LV) function;
    * History of documented congestive heart failure (CHF); and
    * Documented cardiomyopathy
* Uncontrolled hypertension defined as sustained systolic blood pressure (BP) > 150 mmHg or diastolic BP > 90 mmHg; (patients with initial BP elevations are eligible if initiation or adjustment of BP medication lowers pressure to meet entry criteria)
* Active hepatitis B or hepatitis C with abnormal liver function tests
* Intrinsic lung disease resulting in dyspnea
* Poorly controlled diabetes mellitus
* Active infection or chronic infection requiring chronic suppressive antibiotics
* Patients known to be human immunodeficiency virus (HIV) positive with a baseline cluster of differentiation (CD)4 count of < 250 cells/mm^3 or have a history of acquired immune deficiency syndrome (AIDS) indicator conditions; patients taking anti-retroviral therapy that may have a potential overlapping toxicity with the study therapy are not eligible
* Nervous system disorder (paresthesia, peripheral motor neuropathy, or peripheral sensory neuropathy) >= grade 2, per the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0)
* Malabsorption syndrome, ulcerative colitis, resection of the stomach or small bowel, or other disease significantly affecting gastrointestinal function
* Other non-malignant systemic disease that would preclude treatment with any of the treatment regimens or would prevent required follow-up
* Conditions that would prohibit administration of corticosteroids
* Chronic daily treatment with corticosteroids with a dose of >= 10 mg/day methylprednisolone equivalent (excluding inhaled steroids)
* Known hypersensitivity to any of the study drugs or any of the ingredients or excipients of these drugs (e.g., polysorbate 80), including sensitivity to benzyl alcohol
* Pregnancy or lactation at the time of study entry; (note: pregnancy testing must be performed within 2 weeks prior to randomization according to institutional standards for women of childbearing potential)
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements
* Use of any investigational product within 30 days prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2014-02-18 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar F Rimawi, Principal Investigator — NRG Oncology
Locations (732):
- United States (731):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Wilma Chan Highland Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Hematology Oncology Consultants PC-Royal Oak, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Trinitas Hospital and Comprehensive Cancer Center - Williamson Street Campus, Elizabeth, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Newton Medical Center, Newton, New Jersey
  - Chilton Medical Center, Pompton, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Randolph Hospital, Asheboro, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Novant Health Cancer Institute - Rowan, Salisbury, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Winston-Salem Health Care, Winston-Salem, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Surgical Associates Inc, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - Monongalia Hospital, Morgantown, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Ascension Saint Clare's Hospital, Weston, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- San Juan City Hospital, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Combination Chemotherapy, Surgery, Radiation): NEOADJUVANT: Patients receive docetaxel IV over 60 minutes, carboplatin IV over 30-60 minutes, trastuzumab IV over 30-90 minutes, and pertuzumab IV over 30-60 on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients enrolled after Amendment #4 undergo 2 core biopsies prior to course 3 of treatment.
  SURGERY: Patients undergo lumpectomy or mastectomy.
  RADIATION: Patients undergo whole breast irradiation within 8 weeks following surgery.
  ADJUVANT: Patients receive trastuzumab IV over 30-60 minutes every 21 days for up to 1 year.
  Carboplatin: Given IV
  Cytology Specimen Collection Procedure: Undergo 2 core biopsies
  Docetaxel: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pertuzumab: Given IV
  Quality-of-Life Assessment: Ancillary studies
  Therapeutic Conventional Surgery: Undergo lumpectomy or mastectomy
  Trastuzumab: Given IV
  Whole Breast Irradiation: Undergo whole breast irradiation
- Arm II (Chemo, Estrogen Deprivation, Surgery, Radiation): NEOADJUVANT: All patients receive docetaxel, carboplatin, trastuzumab, and pertuzumab as in arm I. Premenopausal patients also receive goserelin acetate SC every 28 days until surgery and aromatase inhibition therapy at the investigator's discretion daily until 1 day before surgery. Postmenopausal patients receive aromatase inhibition therapy at the investigator's discretion daily until 1 day before surgery. Patients enrolled after Amendment #4 undergo 2 core biopsies prior to course 3 of treatment.
  SURGERY: Patients undergo lumpectomy or mastectomy.
  RADIATION: Patients undergo whole breast irradiation within 8 weeks following surgery.
  ADJUVANT: Patients receive trastuzumab IV over 30-60 minutes every 21 days for up to 1 year.
  Aromatase Inhibition Therapy: Given at the investigator's discretion
  Carboplatin: Given IV
  Cytology Specimen Collection Procedure: Undergo 2 core biopsies
  Docetaxel: Given IV
  Goserelin Acetate: Given SC
  Laboratory Biomarker Analysis: Correlative studies
  Pertuzumab: Given IV
  Quality-of-Life Assessment: Ancillary studies
  Therapeutic Conventional Surgery: Undergo lumpectomy or mastectomy
  Trastuzumab: Given IV
  Whole Breast Irradiation: Undergo whole breast irradiation
Period: Overall Study
Arm/Group | Arm I (Combination Chemotherapy, Surgery, Radiation) | Arm II (Chemo, Estrogen Deprivation, Surgery, Radiation)
Started | 158 | 157
Completed | 153 | 155
Not Completed | 5 | 2
Not completed — Patient not at risk for primary endpoint | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Combination Chemotherapy, Surgery, Radiation): Arm I (combination chemotherapy, surgery, radiation)
- Arm II (Chemo, Estrogen Deprivation, Surgery, Radiation): Arm II (chemo, estrogen deprivation, surgery, radiation)
- Total: Total of all reporting groups
Arm/Group | Arm I (Combination Chemotherapy, Surgery, Radiation) | Arm II (Chemo, Estrogen Deprivation, Surgery, Radiation) | Total
Number analyzed (Participants) | 158 | 157 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (11.9) | 50 (10.1) | 50 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 157 | 315
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Pathological Complete Response (pCR) in the Breast and Post Therapy Lymph Nodes
Description: Proportion of patients with pCR evaluated histologically, and defined as the absence of any invasive component in the resected breast specimen and all resected lymph nodes following completion of neoadjuvant therapy.
Time Frame: Up to 2.8 years (when all patients completed primary breast surgery)
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Combination Chemotherapy, Surgery, Radiation) | Arm II (Chemo, Estrogen Deprivation, Surgery, Radiation)
Number analyzed (Participants) | 153 | 155
percentage of participants | 41.2 | 45.8

2. Secondary Outcome: Percent of Patients With Pathologic Complete Response (pCR) in the Breast
Description: Proportion of patients with pCR in the breast, defined as the absence of any invasive component in the resected breast specimen.
Time Frame: Up to 2.8 years (when all patients completed primary breast surgery)
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Combination Chemotherapy, Surgery, Radiation) | Arm II (Chemo, Estrogen Deprivation, Surgery, Radiation)
Number analyzed (Participants) | 153 | 155
percentage of participants | 44.4 | 47.1

3. Secondary Outcome: Recurrence Free Interval (RFI)
Description: Kaplan-Meier estimates of the percentages of patients free from recurrence.
Time Frame: Time from surgery to invasive local, regional or distant recurrence, or death from breast cancer for patients with operable disease and for patients with inoperable progressive disease, assessed up to 8.4 years
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: Overall Survival (OS)
Description: Kaplan-Meier estimates of the percentages of patients surviving.
Time Frame: Time from randomization until death from any cause, assessed up to 8.4 years
Reporting Status: Not Posted, anticipated posting 2025-12

5. Secondary Outcome: Rate of Second Primary Invasive Cancer of Any Type
Description: The cumulative incidence rates of second primary cancers for the two treatment groups.
Time Frame: Time from randomization to the development of a second primary invasive cancer of any site excluding squamous and basal cell carcinoma of the skin, assessed up to 8.4 years
Reporting Status: Not Posted, anticipated posting 2025-12

6. Secondary Outcome: Percent of Patients With Pathological Complete Response (pCR) in the Breast and Post Therapy Lymph Nodes by Menopausal Status
Description: Proportion of patients with pCR evaluated histologically, and defined as the absence of any invasive component in the resected breast specimen and all resected lymph nodes following completion of neoadjuvant therapy calculated separately for premenopausal and postmenopausal women.
Time Frame: Up to 2.8 years (when all patients completed primary breast surgery)
Population: Includes all patients that reported a primary breast cancer surgery.
Measure: Number; unit: percentage of participants with pCR
Arm/Group | Arm I (Combination Chemotherapy, Surgery, Radiation) | Arm II (Chemo, Estrogen Deprivation, Surgery, Radiation)
Number analyzed (Participants) | 153 | 155
percentage of participants with pCR
  Premenopausal Women: number analyzed (Participants) | 77 | 78
  Premenopausal Women | 44.2 | 46.2
  Postmenopausal Women: number analyzed (Participants) | 76 | 77
  Postmenopausal Women | 38.2 | 45.5

7. Secondary Outcome: Patterns of Recurrence Free Interval (RFI) by Menopausal Status
Description: Kaplan -Meier estimates of the percentages of patients free from recurrence by menopausal status.
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: Patterns of Overall Survival (OS) by Menopausal Status
Description: Kaplan-Meier estimates of the percentages of patients surviving by menopausal status.
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2025-12

9. Secondary Outcome: Percentage of Participants With Cardiac Toxicity Categorized According to National Cancer Institute CTCAE Version 4.0
Description: Percentage of patients with grade 1 or higher toxicity from the Cardiac Disorders System Organ Class.
Time Frame: Up to 6 weeks post surgery
Population: Includes all patients that submitted an AE form.
Measure: Number; unit: percentage of pts with cardiac toxicity
Arm/Group | Arm I (Combination Chemotherapy, Surgery, Radiation) | Arm II (Chemo, Estrogen Deprivation, Surgery, Radiation)
Number analyzed (Participants) | 157 | 157
percentage of pts with cardiac toxicity | 4.46 | 4.46

10. Secondary Outcome: Median Percentage of Tumor-infiltrating Lymphocytes (sTILS)
Description: Percentage of Tumor-infiltrating lymphocytes present in the stroma in tissue specimen.
Time Frame: 2.8 years
Population: Includes patients with adequate tissue for assessment of sTILs.
Measure: Median (Inter-Quartile Range); unit: percentage of TILs
Arm/Group | Arm I (Combination Chemotherapy, Surgery, Radiation) | Arm II (Chemo, Estrogen Deprivation, Surgery, Radiation)
Number analyzed (Participants) | 119 | 127
percentage of TILs
  No pCR: number analyzed (Participants) | 73 | 71
  No pCR | 10 [5 to 20] | 10 [0 to 20]
  pCR: number analyzed (Participants) | 46 | 56
  pCR | 10 [5 to 30] | 10 [5 to 22.5]

11. Secondary Outcome: Change in Endocrine-related Symptoms Using Breast Cancer Prevention Trial (BCPT) Symptom Checklist
Description: Mean total score from the BCPT symptom checklist calculated as the average severity score across all items at each timepoint.
Time Frame: Baseline to up to 4 weeks after the last dose of chemotherapy
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an AE form.
Arm/Group | Arm I (Combination Chemotherapy, Surgery, Radiation) | Arm II (Chemo, Estrogen Deprivation, Surgery, Radiation)
Serious Adverse Events (participants affected / at risk) | 36/158 | 35/157
Other Adverse Events (participants affected / at risk) | 151/158 | 151/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Combination Chemotherapy, Surgery, Radiation) (N=158) | Arm II (Chemo, Estrogen Deprivation, Surgery, Radiation) (N=157)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 5 | 6
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bladder infection (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 9 | 5
Diarrhea (Gastrointestinal disorders) | 10 | 13
Dizziness (Nervous system disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 8 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 10 | 6
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Skin infection (Infections and infestations) | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Superficial thrombophlebitis (Vascular disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 1 | 2
Typhlitis (Gastrointestinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 6
Ejection fraction decreased (Investigations) | 1 | 1
Enterocolitis infectious (Infections and infestations) | 3 | 4
Lung infection (Infections and infestations) | 1 | 0
Anorectal infection (Infections and infestations) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Vulval infection (Infections and infestations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Combination Chemotherapy, Surgery, Radiation) (N=158) | Arm II (Chemo, Estrogen Deprivation, Surgery, Radiation) (N=157)
Abdominal pain (Gastrointestinal disorders) | 7 | 12
Alanine aminotransferase increased (ALT/SGPT) (Investigations) | 8 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 66 | 60
Anemia (Blood and lymphatic system disorders) | 75 | 69
Anorexia (Metabolism and nutrition disorders) | 19 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 14
Constipation (Gastrointestinal disorders) | 11 | 7
Creatinine increased (Investigations) | 9 | 5
Dehydration (Metabolism and nutrition disorders) | 47 | 35
Diarrhea (Gastrointestinal disorders) | 93 | 90
Dysgeusia (Nervous system disorders) | 18 | 17
Dyspepsia (Gastrointestinal disorders) | 9 | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 8
Fatigue (General disorders) | 70 | 74
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 13
Headache (Nervous system disorders) | 10 | 11
Hot flashes (Vascular disorders) | 12 | 11
Hyperglycemia (Metabolism and nutrition disorders) | 12 | 10
Hypertension (Vascular disorders) | 26 | 26
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 9
Hypokalemia (Metabolism and nutrition disorders) | 26 | 30
Hypomagnesemia (Metabolism and nutrition disorders) | 10 | 14
Infections and infestations - Other, specify (Infections and infestations) | 7 | 14
Insomnia (Psychiatric disorders) | 13 | 7
Lymphocyte count decreased (Investigations) | 11 | 9
Mucositis oral (Gastrointestinal disorders) | 29 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 12
Nausea (Gastrointestinal disorders) | 61 | 56
Neutrophil count decreased (Investigations) | 22 | 14
Pain (General disorders) | 5 | 17
Peripheral sensory neuropathy (Nervous system disorders) | 16 | 25
Platelet count decreased (Investigations) | 19 | 20
Urinary tract infection (Infections and infestations) | 14 | 19
Vomiting (Gastrointestinal disorders) | 29 | 27
Weight loss (Investigations) | 13 | 13
White blood cell decreased (Investigations) | 11 | 13
Edema limbs (General disorders) | 2 | 11
Ejection fraction decreased (Investigations) | 13 | 6
Infusion related reaction (General disorders) | 3 | 13
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less